CLINICAL TRIAL: NCT05896735
Title: Ultrasound-guided Axillary Vein Catheterization in the Trauma Intensive Care Unit: A Single-Center Retrospective Study
Brief Title: Ultrasound-guided Axillary Vein Catheterization in Trauma
Acronym: UAVCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0364
Record Dates: First submitted 2023-05-02; First posted 2023-06-09 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-04

CONDITIONS: Multiple Trauma/Injuries
Keywords: multiple trauma; axillary vein catheterization; intensive care unit; complications
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ultrasound-guided axillary vein catheterization — All axillary vein catheterizations were performed according to standard central venous catheterization procedures, which were performed under ultrasound guidance at the bedside. Before the operation, patients were placed in a supine position with the upper limb placed in a natural position, and the ultrasound probe and wires were wrapped with a sterile protective sheath. Ultrasound pre-scanning the axillary artery and axillary vein, and pay attention to using the minimum pressure to control the ultrasound probe to avoid crushing the blood vessels. The operator holds the ultrasound probe and puncture needle to puncture the axillary vein under the guidance of ultrasound. After drawing out of the dark red blood, the guide wire was inserted and the puncture needle was withdrawn. The three-lumen CVC catheter was then inserted using the Seldinger technique.

SUMMARY:
It is very important to choose the best central venous catheterization route for trauma patients, the determinants that need to be considered comprehensively include coagulation dysfunction, fracture of the clavicle on the side of the puncture, and tracheotomy care. More importantly, whether it can used simultaneously for accurate volume and invasive hemodynamic monitoring. For the purpose of support of cardiopulmonary function, the ideal position of the catheter tip is vital with regard to an accurate CVP and hemodynamic monitoring. Cannulation of the axillary vein is ideal for patients with severe poly-trauma because it avoids the thoracic cavity, intercostal arteries, tracheostomy, and clavicle, and is prone to compression even if the artery is injured. At present, there is no systematic introduction of ultrasound-guided axillary vein catheterization in the trauma ICU in the literature. Since Oct 2021, the investigators have attempted to practice axillary vein catheterization for this crucial trauma population; unfortunately, the investigators have not know till now whether this procedure is associated with accurate tip placement and its safety should also be weighted. So it is necessary to summarize the relevant clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients admitted to TICU
* Receiving axillary vein catheterization during TICU stay

Exclusion Criteria:

* Without record of axillary vein catheterization
* Without imaging confirming （X-ray or chest CT） the location of catheter tip

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our study do not consider limits on age, sex, or pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Accurate placement of the CVC catheter tip for measuring CVP or invasive hemodynamic monitoring | 2021-10-1~2023-04-30
  Placement of the CVC catheter tip between level of tracheal carina and within 2 cm downward is ideal for measuring CVP or invasive hemodynamic monitoring.

SECONDARY OUTCOMES:
Puncture complications after axillary vein catheterization | 2021-10-1~2023-04-30
  Pneumothorax, thrombus, artery injury, local infection, catheter-related infection
Thromboembolism events | 2021-10-1~2023-04-30
  Incidents of thromboembolism events after axillary vein catheterization during TICU stay
TICU mortality | 2021-10-1~2023-04-30
  Death rate during TICU stay
TICU length of stay | 2021-10-1~2023-04-30
  Time (d) spent during TICU therapy
Ventilator support | 2021-10-1~2023-04-30
  Duration of ventilator support during TICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Shou-Yin Jiang, PhD., Principal Investigator — 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhou J, Wu L, Zhang C, Wang J, Liu Y, Ping L. Ultrasound guided axillary vein catheterization versus subclavian vein cannulation with landmark technique: A PRISMA-compliant systematic review and meta-analysis. Medicine (Baltimore). 2022 Oct 28;101(43):e31509. doi: 10.1097/MD.0000000000031509. PMID 36316830
- [Result] Su Y, Hou JY, Ma GG, Hao GW, Luo JC, Yu SJ, Liu K, Zheng JL, Xue Y, Luo Z, Tu GW. Comparison of the proximal and distal approaches for axillary vein catheterization under ultrasound guidance (PANDA) in cardiac surgery patients susceptible to bleeding: a randomized controlled trial. Ann Intensive Care. 2020 Jul 8;10(1):90. doi: 10.1186/s13613-020-00703-6. PMID 32643012
- [Result] He YZ, Zhong M, Wu W, Song JQ, Zhu DM. A comparison of longitudinal and transverse approaches to ultrasound-guided axillary vein cannulation by experienced operators. J Thorac Dis. 2017 Apr;9(4):1133-1139. doi: 10.21037/jtd.2017.03.137. PMID 28523170
- [Result] Wang HY, Sheng RM, Gao YD, Wang XM, Zhao WB. Ultrasound-guided proximal versus distal axillary vein puncture in elderly patients: A randomized controlled trial. J Vasc Access. 2020 Nov;21(6):854-860. doi: 10.1177/1129729820904866. Epub 2020 Mar 1. PMID 32114875